CLINICAL TRIAL: NCT02450045
Title: Use of Pre-operative Nerve Blocks in Older Patients With Hip Fracture: A Pilot Study
Brief Title: Pre-op Femoral Nerve Block for Hip Fracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00044335
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block (Active Comparator): Patients will receive a pre-operative continuous femoral nerve block.
  Interventions: Procedure: Continuous femoral nerve block; Drug: 0.5% Ropivacaine/0.125% Bupivacaine local anesthetic mixture
- Control (No Intervention): Patients will receive standard care without a continuous femoral nerve block.

INTERVENTIONS:
Procedure: Continuous femoral nerve block
  Arms: Femoral nerve block
Drug: 0.5% Ropivacaine/0.125% Bupivacaine local anesthetic mixture
  Arms: Femoral nerve block

SUMMARY:
Hip fractures (broken hips) are common in older people, particularly older women with fragile bones, and usually occur with a simple fall from a standing height. In Canada, over 28,000 hip fractures occur every year, and approximately 900 occur in Edmonton. After a hip fracture, up to 50% of those who survive their hip fracture do not recover to the same level of activity that they had before breaking their hip. Managing pain with any broken bone is very important. For patients with hip fracture, their older age and fragile health makes pain management even more challenging. Many patients with a hip fracture have reduced ability to think clearly before the fracture. Some patients who have no difficulty with thinking before their hip fracture will become confused for a brief period after their hip fracture or can develop permanent difficulties with thinking. A hip fracture will usually require an operation, and choosing the right pain medication before and after the operation is important since many pain medications make confusion more likely. Permanent difficulty with thinking is a common reason for poor recovery after hip fracture. Our study will look at use of a nerve block to manage pain before patients have their operation. A nerve block provides local pain relief without requiring patients to take the medication by mouth (oral) or through an intravenous (IV) route. A nerve block before surgery may reduce the amount of oral and IV pain medication needed by the patient both before and after their operation but still provide good pain control with less confusion. This could lead to better recovery and allow more patients to return to living in the community rather than long-term care.

DETAILED DESCRIPTION:
Background and rationale

Hip fracture is a common injury in older people, with over 28,000 hip fractures occurring annually in Canada. Approximately 900 hip fractures occur in Edmonton each year. More than 90% of hip fractures result from simple low-energy falls. Many patients who survive do not recover to pre-fracture functional levels and may require permanent long-term care.

The immediate goal of treatment is to control pain while preparing the patient for surgery; greater than 95% of hip fracture patients are treated with surgery to restore mechanical stability and manage pain. Pain after hip fracture has been associated with delirium, depression, sleep disturbance, and decreased recovery. However, in the elderly population, narcotics are also associated with similar side effects such as delirium, cardiovascular and respiratory depression and nausea. This is complicated further in hip fracture patients, in whom pre-existing dementia is common - up to 50% of patients will present with altered cognition. Most studies that examine pain management interventions after hip fracture exclude those with pre-existing dementia. Further research to determine the feasibility of including subjects with cognitive impairment in pain management studies is needed.

Regional anaesthesia can reduce post-operative narcotic use. However, few randomized studies have examined the impact of preoperative regional anesthesia on postoperative outcomes. Effective pain management can affect long-term outcomes: poorly managed pain is associated with delayed ambulation, pulmonary complications, and delayed hospital discharge. Our previous work found limited evidence that nerve blocks may have benefits for hip fracture patients. Other prospective studies have reported the effectiveness of single nerve blocks in reducing narcotic use in Emergency rooms. Continuous preoperative femoral nerve blockade (CFNB) offers the potential benefit of reducing pain in these often frail patients well avoiding adverse outcomes such as delirium. Further work is needed to determine the effectiveness, timing, and safety of a preoperative CFNB on preoperative and postoperative outcomes in the frail hip fracture population, including those with cognitive impairment.

Study objectives

The primary objective is to determine the feasibility of a definitive randomized controlled trial (RCT) that examines the effect of preoperative CFNB in patients with hip fracture, including those with cognitive impairment. Specifically, the investigators will examine 1) Eligibility/recruitment rates; 2) Treatment fidelity; 3) Outcome selection.

The secondary objective is to determine the impact of pre-operative CFNB in patients with hip fracture on the following outcomes within five days of surgery: 1) Proportion of patients with delirium and duration of delirium; 2) Daily pain levels; 3) Total narcotic utilization; 4) Proportion of patients mobilized on postoperative day 1; 4) Readiness for hospital discharge; 5) Complications in hospital, including mortality.

Hypothesis

The investigators hypothesize that pre-operative CFNB will be feasible in this population and will decrease: delirium frequency / duration, pain, and narcotic requirement; will increase the number of patients mobilized on post-operative day 1; and reduce complications and time to readiness for discharge.Study procedures

Research Framework: A complex intervention framework will be used to explore the impact of preoperative CFNB in patients with hip fracture on both preoperative and early postoperative outcomes. The work proposed will undertake initial steps to identify appropriate subjects and assess feasibility and impact of the intervention.

Pilot Study Design: Inception cohort of 75 participants using a concurrent control group with 2:1 allocation of intervention and control subjects. This will allow comparison of outcomes between groups as well as sub-analyses within the intervention group (n=50) to examine treatment fidelity and potential confounding. Although the investigators may be under-powered in this pilot study, they will determine the numbers needed for a future RCT. The proposed sub-analyses will allow us to determine if those with cognitive impairment can be appropriately treated with a CFNB and adequately assessed and if there is an optimal preoperative time frame in which CFNB should be applied.

Intervention: Subjects who score ≥13 on the MMSE, consent to participate, and are recruited within 20 hours of ward presentation will be allocated to receive pre-operative CFNB. Twenty hours was selected as the maximum time that the CFNB could be delayed after presentation to hospital and expect to have an impact on pain management based on anecdotal experience of our Acute Pain Service (APS) team members. The APS will administer the CFNB using a standardized protocol.

Usual Care (Control group): Subjects enrolled after 20 hours of hospital admission (due to delays in obtaining consent) will be allocated to the control group provided that a CAM, required on ward admission as per the hip fracture pathway, was done within 6 hours of ward admission to assess baseline delirium. The investigators do not anticipate selection bias as suitable numbers of patients who are consented before and after 20 hours of admission to the ward should occur.

Femoral Nerve Blockade: The side of hip fracture is identified and marked. With the patient lying supine, the groin is exposed and prepared with 2% chlorhexidine gluconate/70% isopropyl alcohol. A 13-6 MHz high frequency linear ultrasound probe is placed just distal to the lateral edge of the femoral crease and orientated parallel to the crease. The probe is then moved medially, inferior and parallel to the femoral crease, to identify the common femoral artery. The femoral nerve is then identified lateral to the artery and deep to fascia iliaca. Two milliliters of 1% lidocaine is infiltrated subcutaneously at the lateral edge of the probe using a 3 mL syringe and a 25G needle to provide anesthesia to the skin.

A 21G x 95 mm catheter-over-needle assembly is inserted 'in-plane' to the ultrasound probe from the lateral edge of the probe and directed medially under direct visualization to the target position - deep to the fascia iliaca, between the femoral nerve and iliopsoas muscle. The spread of 5 mL dextrose 5% in water injected through the needle confirms correct position. The catheter needle is removed, and the first dose of 20 mL local anesthetic mixture (0.5% Ropivacaine and 0.125% Bupivacaine) is bolused through the catheter using a syringe.

Immediately after, the catheter is secured with a Tegaderm dressing and then connected to an infusion pump programmed to deliver a continuous 1 mL/hr infusion and 4 mL/hr bolus regime of 0.2% Ropivacaine. The infusion/bolus regime is continued until just prior to surgery, at which point, it is discontinued and the catheter bolused with a further 20 mL of local anesthetic mixture prior to catheter removal. Following the regional anesthetic intervention, the subjects are returned to the Orthopaedic ward to await routine surgical care.

Surgery: Surgery within 24-48 hours of admission reduces morbidity and mortality after hip fracture. Over 80% of patients at the UAH are treated within 48 hours of admission. Surgical care will be determined by fracture pattern and patient factors as well perioperative anaesthesia. Study allocation will not affect surgical priority. Both groups will receive routine care pre- and postoperatively as per the clinical pathway, aside from the intervention group receiving the CFNB preoperatively.

Data collection: Baseline data will consist of demographic (e.g., age, gender, residence), medical (cognition (MMSE), delirium (CAM), comorbidities) data and pain using a Visual Analogue Scale (VAS) for those without cognitive impairment and a validated non-verbal pain scale for those with cognitive impairment. Preoperatively, research staff will collect narcotic and non-narcotic analgesic consumption, CAM scores that are performed each shift (i.e., 2 times/day). Pain at rest and with activity will be collected two times/day, between 9-10 am and again between 3-4 pm. During weekend hours, the APS team will collect pain scores. Post-operative data collection will occur until postoperative day 5 or discharge, whichever is sooner. Delirium and pain at rest and with activity will be assessed twice daily as per the preoperative protocol. Narcotic and non-narcotic analgesic utilization will be recorded. The research staff will record when subjects first mobilize (i.e., got up out of bed) and subjects' readiness for discharge (as per the clinical pathway). Complications will also be noted.

Analysis

The process evaluation will assist in determining: 1) Recruitment rate: All patients with hip fracture admitted during the enrollment period will be screened to determine the recruitment rate and generalizability of the cohort; 2) Treatment Fidelity: Defined as delivering the intervention as it was intended, this will be determined by assessing a) the number of Intervention subjects who received the CFNB as prescribed b) the impact of time to CFNB to determine if an optimal preoperative window for the CFNB exists, c) the impact of cognitive impairment on the intervention's effect and the ability to assess outcomes; 3) Outcome Selection: The investigators will evaluate the following issues around outcomes- a) selecting a responsive and appropriate primary outcome measure, b) determining the appropriate time to measure the intervention's impact (i.e., at a single point in time or impact over time), c) comparability of verbal and non-verbal pain assessment, d) completion rate for the clinical pathway elements. The intervention evaluation will determine the impact of preoperative CFNB by comparing outcomes between groups using T-tests and repeated measures analysis of variance (ANOVA) for continuous variables and chi-square tests for categorical variables. Our primary outcome measure for this evaluation will be comparison of delirium between groups using the CAM.

Outcomes

The following standardized outcome measures will be used: Visual Analogue Scale (VAS) for Pain Assessment - Pain at rest and activity will be measured using an 11-point VAS (0-10), a reliable and valid method of measuring patient-reported pain. The Checklist of Non-verbal Pain Indicators (CNPI) has been shown to be reliable and valid in the non-verbal assessment of patients with hip fracture and cognitive impairment. The Confusion Assessment Method (CAM) is able to distinguish between dementia and delirium and can detect delirium in the presence of dementia. Narcotic Consumption - All narcotic medication will be recorded. The total amount of narcotic used will be measured using a morphine equivalency scale with the resulting equivalents totaled to give a single score reflecting the total narcotics used.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory pre-fracture
* Sustained a low-energy hip fracture (i.e., fall from standing)
* Mini Mental Status Examination (MMSE) score of 13 (moderate dementia) or greater
* Consent to participate in study

Exclusion Criteria:

* Failure to obtain consent
* Admitted to hospital more than 30 hours from injury
* Regular use of opiate medications
* Confusion Assessment Method (CAM) test not performed within 6 hours of ward admission
* Known allergy to local anesthetic

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Pain at rest | up to 5 days post-operative
  Visual Analogue Scale and Checklist of Non-verbal Pain Indicators
Pain upon movement | up to 5 days post-operative
  Visual Analogue Scale and Checklist of Non-verbal Pain Indicators

SECONDARY OUTCOMES:
Cognitive function | up to 5 days post-operative
  Confusion Assessment Method
Analgesia consumption | up to 5 days post-operative
  Total narcotic use (morphine equivalency scale)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Beaupre LA, Johnston DB, Dieleman S, Tsui B. Impact of a preemptive multimodal analgesia plus femoral nerve blockade protocol on rehabilitation, hospital length of stay, and postoperative analgesia after primary total knee arthroplasty: a controlled clinical pilot study. ScientificWorldJournal. 2012;2012:273821. doi: 10.1100/2012/273821. Epub 2012 Apr 30. PMID 22666096
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043